CLINICAL TRIAL: NCT02173977
Title: Ultrashort Flare GnRH Agonist Combined With Flexible Multidose GnRH Antagonist Versus Flexible Multidose GnRH Antagonist for Good-prognosis IVF Patients
Brief Title: Ultrashort GnRH Agonist/Antagonist Versus GnRH Antagonist IVF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1078-RO-CTIL
Record Dates: First submitted 2014-06-02; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Infertility
Keywords: GnRH Agonist; GnRH Antagonist; OHSS
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A- Agonist/Antagonist protocol (Active Comparator): The Ultrashort GnRH Agonist/antagonist method entails pre-treatment with oral contraceptive pills before the combination of GnRH ultrashort agonist and antagonist protocol
  Interventions: Other: ARM A- Agonist/Antagonist protocol; Other: ARM B- Antagonist protocol
- ARM B- Antagonist protocol (Active Comparator): The standard IVF method entails Flexible Multidose GnRH Antagonist protocol during COH
  Interventions: Other: ARM A- Agonist/Antagonist protocol; Other: ARM B- Antagonist protocol

INTERVENTIONS:
Other: ARM A- Agonist/Antagonist protocol — In vitro fertilization (IVF/ICSI)
Other: ARM B- Antagonist protocol — In vitro fertilization (IVF/ICSI)

SUMMARY:
The purpose of this study is to evaluate the appropriate controlled ovarian hyperstimulation (COH) protocol in good prognosis patients undergoing IVF treatment. The stimulation characteristics of cycles which include ultrashort flare GnRH agonist combined with flexible multidose GnRH antagonist will be compared to the flexible multidose GnRH antagonist protocol.

The investigators hypothesized that combining the stimulatory effect of GnRH agonists and immediate suppression of the GnRH antagonist in a unique protocol may be a valuable new COH strategy for IVF patients, resulting in improved ART outcome.

DETAILED DESCRIPTION:
The ultrashort flare GnRH agonist combined with flexible multidose GnRH antagonist protocol during COH cycle resulted in a significantly higher clinical pregnancy rate in patients with poor embryo quality, with repeated IVF failures and in poor responders. This protocol combines the effect of the microdose flare on endogenous follicle stimulating hormone (FSH) release with the benefit of an immediate luteinizing hormone suppression of the GnRH antagonist.

The basic hypothesis of this approach can also benefit IVF patients with good prognosis without compromising the ability to use gonadotrophin-releasing hormone (GnRH) agonist to effectively trigger ovulation, while completely eliminating any threat of clinically significant ovarian hyperstimulation syndrome (OHSS).

The purpose of the study is to compare cycles consisting of ultrashort flare GnRH agonist combined with flexible multidose GnRH antagonist with those using the flexible multidose GnRH antagonist protocol

1. To compare the IVF outcome variables and ongoing pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Up to three previous IVF attempts

Exclusion Criteria:

* Patients with poor or no response in previous COH for IVF cycles
* Abnormal ovarian reserve test i.e. anti-mullerian hormone (AMH), Antral follicle test
* Risk factor for Diminished Ovarian Reserve

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | 2 years

SECONDARY OUTCOMES:
Total gonadotropin use | 2 Years
Biochemical pregnancy | 2 Years
  Positive pregnancy test without documentation of intrauterine or extrauterine pregnancy
Clinical pregnancy | 2 Years
  Positive pregnancy test with documentation of intrauterine or extrauterine pregnancy
Multiple pregnancy rate | 2 Years
Miscarriage rate | 2 Years
Fertilization rate | 2 Years
Number of oocytes | 2 years
OHSS rates | 2 Years
Embryo quality | 2 Years
  Grading of a day 3 embryo based on the number of cells that make up the embryo, the amount of fragmentation, and the symmetry of each of the embryo's cells (blastomeres).
  E.g. good quality embryos: embryos that reach the eight-cell stage with less than 20% fragmentation on day 3

OTHER OUTCOMES:
Positive Pregnancy Test | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Orvieto, MD, Principal Investigator — Infertility & IVF Unit, Dept. Obstetrics & Gynecology - Director
Locations (1):
- Sheba Medical Center- IVF unit, Ramat Gan, Israel, Israel

REFERENCES:
- [Background] Orvieto R, Nahum R, Rabinson J, Gemer O, Anteby EY, Meltcer S. Ultrashort flare GnRH agonist combined with flexible multidose GnRH antagonist for patients with repeated IVF failures and poor embryo quality. Fertil Steril. 2009 Apr;91(4 Suppl):1398-400. doi: 10.1016/j.fertnstert.2008.04.064. Epub 2008 Aug 3. PMID 18675974
- [Background] Orvieto R. The ultrashort flare GnRH-agonist/GnRH-antagonist protocol enables cycle programming and may overcome the "detrimental effect" of the oral contraceptive. Fertil Steril. 2012 Sep;98(3):e17-8; author reply e19. doi: 10.1016/j.fertnstert.2012.06.053. Epub 2012 Jul 26. No abstract available. PMID 22840381
- [Background] Orvieto R, Nahum R, Zohav E, Liberty G, Anteby EY, Meltcer S. GnRH-agonist ovulation trigger in patients undergoing controlled ovarian hyperstimulation for IVF with ultrashort flare GnRH-agonist combined with multidose GnRH-antagonist protocol. Gynecol Endocrinol. 2013 Jan;29(1):51-3. doi: 10.3109/09513590.2012.705376. Epub 2012 Aug 3. PMID 22857268
- [Background] Orvieto R, Meltcer S, Liberty G, Rabinson J, Anteby EY, Nahum R. A combined approach to patients with repeated IVF failures. Fertil Steril. 2010 Nov;94(6):2462-4. doi: 10.1016/j.fertnstert.2010.03.057. Epub 2010 May 7. PMID 20451192
- [Background] Orvieto R, Kruchkovich J, Rabinson J, Zohav E, Anteby EY, Meltcer S. Ultrashort gonadotropin-releasing hormone agonist combined with flexible multidose gonadotropin-releasing hormone antagonist for poor responders in in vitro fertilization/embryo transfer programs. Fertil Steril. 2008 Jul;90(1):228-30. doi: 10.1016/j.fertnstert.2007.06.022. Epub 2007 Aug 6. PMID 17681292